CLINICAL TRIAL: NCT04939246
Title: A Feasibility Study of Stereotactic MRI-guided Adaptive Radiation Therapy (SMART) in One Fraction for Inoperable Primary or Metastatic Carcinoma (SMART ONE)
Brief Title: Stereotactic MRI-guided Adaptive Radiation Therapy (SMART) in One Fraction
Acronym: SMART ONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baptist Health South Florida (Other)
Collaborators: Viewray Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-CHU-002
Record Dates: First submitted 2021-06-10; First posted 2021-06-25 (Actual); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Carcinoma
MeSH Terms: conditions — Carcinoma | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single-fraction SABR (Other): Patients will receive SABR in a single-fraction regiment treatment with one single dose of radiation therapy per lesion. Patients may be treated for up to a total of ten lesions. Each lesion will be treated in one fraction.
  Interventions: Radiation: Stereotactic ablative body radiation therapy

INTERVENTIONS:
Radiation: Stereotactic ablative body radiation therapy — Single-fraction of stereotactic ablative body radiation (SABR) therapy will be delivered with an integrated magnetic resonance imaging (MRI)-guided radiotherapy delivery system (ViewRay MRIdian Linac). The prescription dose is dependent on the anatomic location of the lesion and based on previously published safety data.

SUMMARY:
This is a multi-site single arm feasibility study of single-fraction Stereotactic MRI-guided Adaptive Radiation Therapy (SMART) for primary or metastatic carcinoma involving the lung, liver, adrenal gland, abdominal/pelvic lymph node, pancreas, and/or kidney. Stereotactic ablative body radiation therapy (SABR) is a highly-focused radiation treatment that gives an intense dose of radiation concentrated on a tumor, while limiting the dose to the surrounding organs.

ELIGIBILITY:
Inclusion Criteria

1. Subject must be ≥18 years of age at the time of study enrollment
2. Subject must have Biopsy-confirmed primary or metastatic carcinoma with involvement of the lung, liver, adrenal gland, pancreas, kidney, and/or abdominal/pelvic lymph node that would receive SABR
3. Any lesion that would receive SABR under this study protocol is no larger than 5 cm in greatest dimension
4. 1-10 total lesions that would receive SABR
5. If multiple lesions are treated, they must be at least 3 cm apart
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
7. Life expectancy at least 6 months
8. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Abstinence is acceptable if it's the patient preferred method. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
9. Patients receiving hormonal therapy or immunotherapy such as immune checkpoint inhibitor that had begun at least 4 weeks prior to SABR will be allowed.

Exclusion criteria

1. Subject has contraindication to having an MRI scan
2. Subject has central or ultra-central lung tumor that would receive SABR on this study, defined as a lesion located within 2 cm of the trachea and proximal bronchial tree
3. Subject has received cytotoxic chemotherapy or investigational agent within 2 weeks of SBRT
4. Subject has uncontrolled brain metastases, spinal cord compression, or leptomeningeal carcinomatosis
5. Subject has any unresolved toxicity (Common Terminology Criteria for Adverse Events version 5.0 > grade 2) from previous anti-cancer therapy
6. Subject has any condition in the opinion of the investigator that would interfere with evaluation of study treatment or interpretation of patient safety or study results
7. Subject has received prior radiation therapy that directly overlaps any radiation therapy given in this study
8. Subject has received radiation therapy that could lead to an unacceptably high risk of clinically significant normal tissue injury due to high cumulative normal tissue dose as determined by the investigator
9. Female subject who are pregnant or breastfeeding
10. Subject who has received vascular endothelial growth factor (VEGF) inhibitor such as bevacizumab within 4 weeks prior to study therapy or planned to receive it within 4 weeks after study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Chuong, MD, Principal Investigator — Miami Cancer Institute (MCI) at Baptist Health, Inc.
Locations (2):
- United States (2):
  - Miami Cancer Institute at Baptist Health South Florida, Miami, Florida
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chuong MD, Mittauer KE, Bassetti MF, Rojas C, Glide-Hurst C, Kalman NS, Tom MC, Rubens M, Crosby J, Burr A, Tolakanahalli R, Gutierrez AN, Bassiri N, Mehta MP, Kotecha R. Stereotactic Magnetic Resonance Guided Adaptive Radiation Therapy in One Fraction (SMART ONE): A Multicenter, Single-Arm, Phase 2 Trial. Int J Radiat Oncol Biol Phys. 2025 Jul 15;122(4):957-967. doi: 10.1016/j.ijrobp.2025.03.030. Epub 2025 Mar 28. PMID 40158734
- See also: MCI - Website — http://baptisthealth.net/cancer-care/home

RESULTS

PARTICIPANT FLOW:
Period: Screening
Arm/Group | Single-fraction SABR
Started | 30
Completed | 30
Not Completed | 0
Period: During Treatment
Arm/Group | Single-fraction SABR
Started | 30
Completed | 30
Not Completed | 0
Period: After Treatment
Arm/Group | Single-fraction SABR
Started | 30
Completed | 23
Not Completed | 7
Not completed — Death | 4
Not completed — Lost to Follow-up | 1
Not completed — Discharged to hospice | 2

BASELINE CHARACTERISTICS:
Units Other Than Participants: lesions
Arm/Group | Single-fraction SABR
Number analyzed (Participants) | 30
Number analyzed (lesions) | 32
Age, Continuous [Median (Full Range); unit: years] | 69 [49 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — ECOG describes a participant's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). It is assessed on a scale of 0 (fully active) to 5 (dead). Participants must have had a baseline score of 0 to 2 to be considered eligible for this study.
  participants
    0 (Fully active, able to carry on all pre-disease performance without restriction) | 12
    1 (Ambulatory, able to carry out work of a light or sedentary nature) | 18
Previous Systemic Therapy for Metastatic Disease [Number; unit: participants]
  Chemotherapy Only | 10
  Immunotherapy Only | 2
  Chemotherapy and Immunotherapy | 2
  None | 16
Total Number of Treated Lesions [Number; unit: lesions] | 32
Maximum Size of Treated Lesions [Median (Full Range); unit: cm] | 1.7 [1.0 to 3.9]
Primary or Metastatic Lesions [Number; unit: lesions]
  Primary | 2
  Metastatic | 30
Anatomic Location [Number; unit: lesions]
  Lung | 11
  Adrenal gland | 9
  Abdominal/pelvic lymph node | 6
  Liver | 5
  Pancreas | 1
Primary Tumor Location [Number; unit: lesions]
  Colon/rectum | 16
  Lung | 10
  Kidney | 2
  Esophagus | 1
  Pancreas | 1
  Anal canal | 1
  Tonsil | 1
Primary Tumor Definitively Managed [Count of Participants; unit: Participants]
  Yes | 27
  No | 1
  Not Applicable | 2
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 17
  Non-small cell lung carcinoma | 7
  Squamous cell carcinoma | 3
  Renal cell carcinoma | 2
  Small cell lung carcinoma | 1
Interval from Initial Diagnosis to Enrolment [Median (Full Range); unit: months] | 20.1 [1.9 to 79.0]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With SABR Successfully Delivered in One Fraction
Description: To be considered successful, SABR treatment must meet the following criteria:
  1. Successful completion of treatment to each lesion within 3 days of intended treatment date
  2. Successful completion of treatment to each lesion within 90 minutes from the patient entering the treatment room until treatment completion for at least 80% of treated lesions
  3. Image guidance verification of treatment delivery within 5 mm of the planned delivery
Time Frame: through study completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Single-fraction SABR
Number analyzed (Participants) | 30
Participants | 30

2. Primary Outcome: Number of Patients Demonstrating Tolerability
Description: Number of patients that meet the following criteria:
  1. No greater than 4 of 30 patients experience grade 3 or higher acute toxicity is attributable to SABR within 90 days of completing SABR
  2. No grade 5 toxicity is attributed to SABR
Time Frame: through study completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Single-fraction SABR
Number analyzed (Participants) | 30
Participants
  Did not meet toxicity criteria | 28
  Grade 3 or higher acute toxicity attributable to SABR (excludes Grade 5 toxicities in next category) | 2
  Grade 5 toxicity attributed to SABR | 0

3. Secondary Outcome: One-year Local Control
Description: Assessed using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and estimated with Kaplan-Meier and corresponding 95% confidence interval from the time of study treatment.
  Target lesion:
  * Complete response (CR): Disappearance of all target lesions
  * Partial response (PR): >30% decrease in the sum of the diameters of target lesions
  * Stable disease (SD): Target lesion has neither sufficient decrease to qualify as a PR or sufficient increase to qualify as progressive disease (PD)
  * PD: At least a 20% increase in the sum of the diameters of target lesions an absolute increase of at least 5 mm
  Non-target lesion:
  * CR: Disappearance of all non-target lesions
  * SD: Persistence of ≥1 non-target lesions
  * PD: Appearance of ≥1 new lesions or unequivocal progression of existing non-target lesions
  Overall:
  * CR: Target CR+non-target CR
  * PR: Target CR/PR+non-target non-PD
  * SD: Target SD+non-target non-PD
  * PD: Anything else
  Local control=CR+PR+SD using overall response.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single-fraction SABR
Number analyzed (Participants) | 30
percentage of participants | 96.2 [88.8 to 100.00]

4. Secondary Outcome: Percent of Participants With One-year Overall Survival
Description: Percent of participants with one-year overall survival will be estimated using the Kaplan-Meier method along with the corresponding 95% confidence interval from the time of study treatment.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single-fraction SABR
Number analyzed (Participants) | 30
percentage of participants | 86.3 [73.8 to 98.8]

5. Secondary Outcome: Number of Participants With Acute and Late Toxicity Results
Description: Number of participants with acute and late toxicities defined as grade 3 or higher toxicity attributable to SABR will be determined. For patients receiving SABR to multiple lesions, acute toxicity will be determined from the date of the initiation of SABR.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Single-fraction SABR
Number analyzed (Participants) | 30
participants
  Acute | 2
  Late | 0

6. Secondary Outcome: Change in Participant Reported Quality of Life Questionnaire
Description: Patient-reported quality of life will be determined using the Functional Assessment of Cancer Therapy - General (FACT-G) survey instrument. FACT-G is a 27-item questionnaire that covers four sub-domains: physical (7 items), social (7 items), emotional, (6 items), and functional (7 items) well-being. Each question is scored from a scale from 0 (not at all) to 4 (very much) using a manual scoring template in which some items are reversed. After reversal of specified items, the sub-domain scores are totaled, then multiplied by the number of items in the sub-domain, and then divided by the number of items the participant answered. The scores for each sub-domain are 0 (worst well-being) to 24 (best emotional well-being) or 28 (best physical, social, or functional well-being). The total scores can range from 0 (worst overall well-being) to 108 (best overall well-being).
Time Frame: baseline, 3, 6, 9, and 12 months after treatment
Measure: Median (Full Range); unit: score on a scale (FACT-G)
Arm/Group | Single-fraction SABR
Number analyzed (Participants) | 30
score on a scale (FACT-G)
  Baseline | 84 [29.2 to 112]
  3 Months | 85 [56 to 104]
  6 Months | 69 [0 to 104]
  9 Months | 91 [0 to 108]
  12 Months | 93 [65.2 to 108]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Single-fraction SABR
All-Cause Mortality (participants affected / at risk) | 4/30
Serious Adverse Events (participants affected / at risk) | 3/30
Other Adverse Events (participants affected / at risk) | 28/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-fraction SABR (N=30)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-fraction SABR (N=30)
Fatigue (General disorders) | 12 (13)
Abdominal Pain (Gastrointestinal disorders) | 9 (9)
Nausea (Gastrointestinal disorders) | 5 (7)
Anemia (Blood and lymphatic system disorders) | 4 (5)
Hypertension (Vascular disorders) | 4 (4)
Creatinine Increased (Investigations) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Urinary Tract infection (Infections and infestations) | 2 (3)
Alkaline phosphatase increased (Investigations) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Lymphocyte count decreased (Investigations) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Investigations, Other - Platelet count increased (Investigations) | 2 (2)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/46/NCT04939246/Prot_SAP_000.pdf